CLINICAL TRIAL: NCT05760664
Title: Exercises Directed To Dynamic Stiffness Of The Thoracolumbar Region And Performance Of Amateur Runners: Randomized Controlled Clinical Trial
Brief Title: Exercises Directed To Dynamic Stiffness Of The Thoracolumbar Region And Performance Of Amateur Runners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Principal Investigator, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dynamic Stiffness of runners
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Fascia
Keywords: Sports Performance; Fascia; Running
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): The fascial fitness® method (12 sessions, twice a week, for six weeks, 15 minutes a day, for 2 sets of 40 seconds each side). Assessments and reassessments will be carried out in the first, fourth and sixth week.
  Interventions: Other: Group Experimental/Fascial Fitness
- Sham Group (Active Comparator): Static stretching exercises (12 sessions, twice a week, for six weeks, 15 minutes a day, for 2 sets of 40 seconds each side). Assessments and reassessments will be carried out in the first, fourth and sixth week.
  Interventions: Other: Group Sham/Static stretching exercise
- Control Group (Placebo Comparator): The placebo intervention will be performed using ultrasound turned off in the thoracolumbar region for 15 minutes followed by rest for 15 minutes for 6 weeks, twice a week. Ultrasound was chosen because it is easy-to-use equipment and because this form of placebo used, equipment turned off, does not have any treatment effect and has already been established in another study (CHAIBI; BENTH; RUSSELL, 2015). Assessments and reassessments will be carried out in the first, fourth and sixth week.
  Interventions: Other: Control Group/Placebo

INTERVENTIONS:
Other: Group Experimental/Fascial Fitness — Participants will receive twelve treatment sessions, twice a week, for six weeks, lasting 30 minutes per session. The interventions will be applied by a physiotherapist with previous experience and training in the proposed protocols.
  Arms: Experimental Group
Other: Group Sham/Static stretching exercise — Participants will receive twelve treatment sessions, twice a week, for six weeks, lasting 30 minutes per session. The interventions will be applied by a physiotherapist with previous experience and training in the proposed protocols.
  Arms: Sham Group
Other: Control Group/Placebo — The placebo intervention will be performed using ultrasound turned off in the thoracolumbar region for 15 minutes followed by rest for 15 minutes for 6 weeks, twice a week. Participants will be evaluated on the first day, fourth week and sixth week of intervention.
  Arms: Control Group

SUMMARY:
Introduction: Worldwide, the number of amateurs runners is growing exponentially, with consequent increase in musculoskeletal injuries. Although prevention and treatment by myofascial release has shown some evidence over the years, many issues remain. However, this evidence is based on studies that are not randomized controlled trials. Thus, issues associated with prevention and treatment strategies and their effects have not yet been fully explored by researchers. Objective: Contribute to the formation of basic knowledge and understanding of the impact of exercises aimed at the fascial system (fascial fitness®) on the dynamic stiffness of the thoracolumbar region and on the performance of amateur runners. Methods: This project tests a randomized, double-blind (evaluator and patient), parallel clinical trial in three groups comparing the effects of fascial fitness®, kinesiotherapy and placebo for a dynamic stiffness of the thoracolumbar thoracolumbar region and for the performance of amateur runners. Participants will be randomly allocated to receive a 6-week fascial fitness® program, either kinesiotherapy or placebo (detuned ultrasound). Outcome measures will be used before interventions, 3 and 6 weeks after randomization. Interventions will be cared out twice a week for six weeks. Primary outcomes will be the dynamic stiffness of the thoracolumbar region and the time to complete the 5 km run. As secondary outcomes form the ability to maintain static posture in three different postures, the pressure pain threshold, the electromyographic activity of the latissimus dorsi muscle, the quality of movement patterns and heart rate variability in the 5 km run. To analyze whether fascial fitness® or kinesiotherapy or placebo will mediate changes in outcome variables, multivariate analysis of variation will be used.

ELIGIBILITY:
Inclusion Criteria:

Eligible runners must meet the following criteria:

* 5km amateur runners;
* 18 to 45 years old;
* the both sexes;
* be performing running activity for at least 1 year;
* training rate of at least twice a week.

Exclusion Criteria:

* Difficulty in understanding the Portuguese language to answer the questionnaires;
* self-report of carrying neuromusculoskeletal diseases;
* trauma or surgeries in the last 90 days in the lower limbs;
* vestibular system in the last 30 days;
* controlled medicine;
* previous physiotherapeutic treatment in the last 30 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic stiffness | 6 weeks
  The primary outcomes will be the dynamic stiffness of the thoracolumbar region and the time to run 5 km. Muscle stiffness will be measured in a relaxed state using a portable device, the MyotonPRO (Myoton AS, Tallinn, Estônia), which applies a short (15 ms) mechanical impulse to cause damped oscillations in the muscle.

SECONDARY OUTCOMES:
Pressure pain threshold | 6 weeks
  For the evaluation of the pressure pain threshold, the participant will be in ventral decubitus with the algebrameter positioned perpendicular to the region of two fingers laterally to the spinous process of L4, in the latissimus muscle of the back of the predominant side. The evaluator will perform pressure perpendicular to the skin up to the maximum pain tolerance supported by the subject and reported by the subject twice, and the mean value between the two measurements will be used.
Functional Moviment Screen | 6 weeks
  The quality of the movement patterns will be evaluated by the Functional Moviment Screen. Seven postures will be applied: Deep Squat (deep squat that evaluates bilaterally and symmetrically, the functionality of the hips, knees and ankles), Hurdle Step (one step through an obstacle, examining the mechanics of the stride), In line Lunge (hip and trunk mobility, ankle and knee stability, and hamstring flexibility), Shoulder Mobility (shoulder mobility bilaterally), Active Straight-Leg Raise (actively lift the leg in knee extension, determining tendon activity and flexibility of gastrocnemius-sumour, while maintaining a stable pelvis), Trunk Stability Push-up (trunk stability, while upper-member symmetry is performed) and Rotary Stability (rotation stability test, which assesses trunk stability while upper and lower limbs are in combined motion).
Vertical Jump | 6 weeks
  The vertical jump assessment will be performed with the individual with their hands on their hips, from a static position and with their legs straight during the entire jump phase, the landing must be performed with both feet, keeping the ankles dorsiflexed .

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil